CLINICAL TRIAL: NCT06229925
Title: Effects of Transcranial Direct Current Stimulation Versus Sham in Subacromial Pain Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Transcranial Direct Current Stimulation Versus Sham in Subacromial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor and Researcher, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VDS2024
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Subacromial Pain Syndrome; Transcranial Direct Current Stimulation
Keywords: Transcranial Direct Current Stimulation; Neuromodulation; Pain in the shoulder; Chronic pain; Treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Stimulation (Experimental): Active direct current stimulation for 20 minutes.
  Interventions: Device: Experimental Stimulation
- Sham Stimulation (Sham Comparator): Sham direct current stimulation for 20 minutes.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Experimental Stimulation — Application of active direct current stimulation for 20 minutes, at an intensity of 2mA, with 30s of ramp up and ramp down, for 5 consecutive days. The anode will be positioned on M1 (C3) contralateral to the painful shoulder; The reference electrode (cathode) will be placed in the supraorbital region contralateral to the anode (Fp2). Direct current will be delivered through two 35cm2 surface sponge electrodes (7x5) soaked in saline solution, using a portable neuromodulator. During the entire stimulation, volunteers will remain seated in an air-conditioned and quiet place.
  Arms: Experimental Stimulation
Device: Sham Stimulation — Application of active direct current stimulation for 20 minutes, at an intensity of 2mA, for 5 consecutive days, administered in the same way as the experimental intervention. However, the stimulator will be turned off after 30 seconds and the volunteers will not receive current for the rest of the session.
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to investigate the effects of applying Transcranial direct current stimulation on pain levels and function, quality of life, muscle strength and range of motion in individuals with subacromial pain syndrome.

DETAILED DESCRIPTION:
This is a controlled, randomized and blind clinical trial, which will be carried out with individuals from the city of Natal/RN, aged between 18 and 65 years, of both sexes, diagnosed with subacromial pain syndrome, who present a level of pain greater than 3 on the Numerical Pain Scale, at rest, for at least 3 months. The research sample will be non-probabilistic, in which they will be randomly distributed into two distinct groups: active tDCS (active stimulation) and sham tDCS (stimulation turned off after 20 seconds). This research was submitted to the UFRN Research Ethics Committee through the national interface Plataforma Brasil. This research covers the ethical aspects guided by Resolution 466/2012 of the National Health Council and the Declaration of Helsinki for research with human beings. In addition, the research will be registered in Clinical Trials. All data will be recorded in the laboratory's database under confidentiality and may only be processed by the responsible researchers. The study will only begin after the issuance of the reference opinion approving the project. All subjects will be duly informed and guided regarding the scheduled procedures, which will only be carried out after reading, accepting and signing the Informed Consent Form. After approval by the Research Ethics Committee, following resolution 466/2012, a pilot study was carried out to adapt all research procedures, as well as training the researchers involved. Volunteers will be duly informed about the objectives and advantages of their participation in the study, and will then undergo an assessment of pain sensation, using the Numerical Pain Scale; assessment of shoulder range of motion, using the Smartphone clinometer application; assessment of muscle strength through flexion, hyperextension, medial and lateral rotation movements of the shoulder, using a portable dynamometer; will complete the Douleur Neuropathique 4 questionnaire (DN4) to screen for neuropathic pain, the Disabilities of the arm, shoulder and hand questionnaire (DASH) to assess upper limb function, and the Short Form 36 Health Survey questionnaire (SF-36) to assess health-related quality of life. They will then undergo 20 minutes of stimulation for 5 consecutive days, according to the pre-determined group. The assessments will be repeated at the end of the intervention and in a 1-week follow-up, in which they will receive an educational booklet.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral pain in one shoulder
* Pain level ≥ 3 on the Numerical Pain Scale (END), at rest, for at least 3 months
* No previous treatment with tDCS
* Present graded disability on the DASH questionnaire (> 15 points)
* At least three positive tests, among the five indicated below: Neer, Hawkins, Jobe, Patte or painful abduction arch.

Exclusion Criteria:

* Indication for surgical repair and/or history of shoulder surgery
* Shoulder fracture and/or dislocation
* Partial or total rupture of one of the rotator cuff tendons and/or the long head of the biceps
* Fibromyalgia
* History of epilepsy
* Panic syndrome
* Implantable devices in the skull
* Significant neurological or psychiatric diseases
* Severe cardiopulmonary, renal and hepatic diseases
* Current pregnancy.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (numerical pain rating scale) | Up to 1 week of follow-up
  Pain intensity measured by numerical pain rating scale, measured on an 11-point where 0=no pain and 10=worst possible pain.

SECONDARY OUTCOMES:
Peak of muscular torque | Up to 1 week of follow-up
  Evaluate the peak of muscular torque using the hand-held dynamometer.
Range of motion (ROM) | Up to 1 week of follow-up
  Evaluate the range of motion using the Smartphone clinometer application
Degree of disability of the upper limbs | Up to 1 week of follow-up
  Evaluate the degree of disability of the upper limbs using the Disabilities of the arm, shoulder and hand (DASH) questionnaire. Total scores range from 0 to 100 for each dimension, with higher values indicating worse upper limb function.
Health-related Quality of Life | Up to 1 week of follow-up
  Evaluate the health-related Quality of Life using the Quality of Life questionnaire (SF-36). The score for this questionnaire ranges from 0 to 100, with higher values indicating a better general state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Vinícius Dantas, Esp, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No